CLINICAL TRIAL: NCT03489135
Title: The Venous Thrombus Extraction (VETEX) Clinical Study: A Preliminary Investigation
Acronym: VETEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vetex Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VETEX
Record Dates: First submitted 2018-03-28; First posted 2018-04-05 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Deep Vein Thrombosis Leg
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention using the ReVene Thrombectomy Catheter (Experimental): Open label, prospective, non-randomised, multi-centre first-in-human evaluation of the Vetex ReVene Thrombectomy Catheter for treatment of acute iliofemoral deep vein thrombosis (DVT).
  Interventions: Device: ReVene Thrombectomy Catheter

INTERVENTIONS:
Device: ReVene Thrombectomy Catheter — Endovascular treatment of an acute iliofemoral DVT

SUMMARY:
This is an open label, prospective, non-randomised, multi-centre first-in-human evaluation of the Vetex Thrombectomy Device for treatment of acute iliofemoral deep vein thrombosis (DVT)

ELIGIBILITY:
Inclusion Criteria:

1. Men and women over 18 years of age
2. Unilateral Iliofemoral DVT
3. Patients with acute iliofemoral DVT confirmed by imaging Colour Doppler Ultrasonography (CDUS) and Magnetic Resonance Venography (MRV) or CT Venography (CTV) with symptom duration not exceeding 14 days at presentation
4. Voluntary written consent, given before performance of any clinical investigation-related procedure not part of standard medical care, and with the understanding that consent may be withdrawn at any time without prejudice to future medical care.
5. Female subjects must also meet any one of the following criteria:

   1. Surgically sterile with bilateral tubal ligation or hysterectomy
   2. Post-menopausal for at least one year
   3. If of child-bearing potential, a pregnancy test should be performed and they should be practicing an acceptable method of birth control for the duration of the clinical investigation as judged by the Investigator, such as condoms, foams, jellies, diaphragm, intrauterine device or abstinence.
6. Subjects willing to undergo pre-and post-clinical investigation blood and urine investigations.
7. Good Functional Status as determined by the physician

Exclusion Criteria:

1. Age less than 18 years
2. Symptom duration > 14 days for the DVT episode in the index leg (i.e., non-acute DVT)
3. Inferior Vena Cava (IVC) Atresia
4. Previously stented in treatment vein
5. Patients with Antiphospholipid Syndrome
6. In the index leg: established Post-Thrombotic Syndrome (PTS)
7. Bilateral disease
8. Limb-threatening circulatory compromise
9. Known symptomatic Pulmonary Embolism
10. Hemodynamically compromised (i.e., hypotension).
11. Patients with severe dyspnea or acute systemic illness.
12. Allergy, hypersensitivity, or thrombocytopenia from heparin, rt-PA, or iodinated contrast, except for mild-moderate contrast allergies for which steroid pre-medication can be used.
13. Hemoglobin < 9.0 mg/dl, INR > 1.6 before warfarin was started, or platelets < 100,000/ml.
14. Impaired renal function (estimated glomerular filtration rate (GFR) < 30 ml/min), defined as serum creatinine ≥133µmol/L for male and ≥125 µmol/L for female.
15. Active bleeding, recent (< 3 months) gastrointestinal (GI) bleeding, severe liver dysfunction, bleeding diathesis.
16. Recent (< 3 months) internal eye surgery or hemorrhagic retinopathy; recent (< 10 days) major surgery, cataract surgery, trauma, cardiopulmonary resuscitation (CPR), obstetrical delivery, or other invasive procedure.
17. History of stroke or intracranial/intraspinal bleed, tumor, vascular malformation, aneurysm.
18. Active cancer (metastatic, progressive, or treated within the last 6 months). Exception: patients with non-melanoma primary skin cancers are eligible to participate in the study.
19. Severe hypertension on repeated readings (systolic > 180 mmHg or diastolic > 105 mmHg).
20. Pregnant (positive pregnancy test, women of childbearing potential must be tested).
21. Recently (< 1 month) had thrombolysis
22. Life expectancy < 1 year or chronic non-ambulatory status.
23. Participation in any other device study within the last year, which has not yet met the primary endpoint.
24. Patient has any concurrent condition that, in the Investigator's opinion, would jeopardize the safety of the subject or compliance with the protocol.
25. Likely inability to comply with the protocol or cooperate fully with the investigator and site personnel.
26. Impaired liver function, defined as ALT or AST ≥2.5 times upper normal limit (UNL).
27. Clinically significant, active disease (within 12 months) of the pulmonary, gastrointestinal, neurological, genitourinary or haematological system, that in the opinion of the Investigator, may confound the results of the trial or pose additional risk to the subject following use of the Vetex Thrombectomy Device.
28. Cardiac disorder, defined as: congestive heart failure (New York Heart Association (NYHA) class III/IV), diagnosis of unstable angina pectoris, cerebral stroke and or myocardial infarction within the last 12 months or planned coronary or carotid revascularisation procedures.
29. Atrial/Ventricular Septal Defect
30. Mental incapacity, unwillingness or language barrier precluding adequate understanding of the trial procedure or cooperation with trial site personnel.
31. Known or suspected abuse of alcohol, narcotics or non-prescription drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Primary Performance Outcome | 0 days
  • Procedural success, defined as successful preparation and use of the device to achieve Society Interventional Radiology (SIR) Grade II Lysis (50-95% thrombus removal) in the target vessel, with freedom from procedural related adverse events

CONTACTS AND LOCATIONS:
Locations (5):
- Bulgaria (2):
  - City Clinic Burgas, Burgas
  - City Clinic Sofia, Sofia
- Klinikum Hochsauerland GmbH, Arnsberg, Germany
- University Hospital Galway, Galway, Ireland
- Guys and St. Thomas, London, United Kingdom